CLINICAL TRIAL: NCT04732078
Title: Physical and Mental Characteristics in Active Elderly People and Their Influence on Quality of Life
Brief Title: Physical and Mental Characteristics in Active Elderly People
Acronym: ActivOld
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Other Study IDs: ID0032
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Old Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today's world is characterized among other things by a progressive increase in the aging population, due to a decrease in the birth rate and an increase in life expectancy. In developed countries, the number of older people is increasing, largely due to significant advances in health sciences and new life habits. The aim of this study is to describe an active population over 60 years old, which complies with the concept of successful aging, in order to know its characteristics both at a physical and mental health level and to be able to make recommendations from physiotherapy. Active people over 60 years of age recruited from two associations (Amics de la Nau Gran, and Hogares) from the city of Valencia, Spain will be part of the study.

Pain was assessed using the Visual Analogue Scale, the level of physical activity performed using the IPAQ questionnaire, quality of life using the SF-12v2, sleep quality using the Pittsburg questionnaire, and mood using the depression scale and Goldberg's anxiety, as well as functional tests to assess respiratory status.

DETAILED DESCRIPTION:
Today's world is characterized among other things by a progressive increase in the aging population, due to a decrease in the birth rate and an increase in life expectancy. In developed countries, the number of older people is increasing, largely due to significant advances in health sciences and new life habits. The practice of physical activity is rapidly becoming a constant among the population (as its many health benefits are becoming known) and increasingly among the elderly population. As there are no previous studies in our country that observe and relate different physical and mental aspects in older active population that complies with the concept of "successful aging", it has been decided to carry out this research to try to detect the benefits and deficiencies present in the condition health of people considered active and over 65 years. From the results obtained, recommendation strategies from physiotherapy can be defined and the effects that the practice of physical activity has on different aspects of the person's health will be shown. Our hypothesis of the present study is that active older people who frequently engage in physical activity have good mental and physical health, as well as good respiratory condition and quality of life.

Objective: Describe an active population over 60 years old, which complies with the concept of successful aging, in order to know its characteristics both at a physical and mental health level and to be able to make recommendations from physiotherapy.

In addition, analyze the state and the different respiratory variables in an active elderly population, know the state of mental health, detect signs related to anxiety or depression, know the quality and possible sleep disorders. Also analyze and relate physical health and mental health, and know the level of quality of life in this population group.

Material and methods Study design. Descriptive study developed at the University of Valencia. Participants. Active people over 60 years of age recruited from two associations from the city of Valencia, Spain will be part of the study.

Pain was assessed using the Visual Analogue Scale, the level of physical activity performed using the IPAQ questionnaire, quality of life using the SF-12v2, sleep quality using the Pittsburg questionnaire, and mood using the depression scale and Goldberg's anxiety, as well as functional tests to assess respiratory status.

ELIGIBILITY:
Inclusion Criteria:

* That they obtain in the IPAQ questionnaire on physical activity values belonging to category 2 (moderate level of physical activity) or 3 (high level of physical activity), that is, belonging to the group of ACTIVE people.
* That they are suitable in the Lobo Mini Cognitive Exam, with a score greater than or equal to 24 (with an adequate level of cognition, necessary to carry out the study).
* Meet the characteristics of "successful aging" (not having suffered in the last two years stroke or cerebrovascular accident, arteriosclerosis, angina, acute myocardial infarction, cancer, diabetes, chronic respiratory disease, chronic cardiovascular disease, neurological disease or psychological alteration).

Exclusion Criteria:

* Under 60 years not active according to the IPAQ
* Score less than 24 in the Lobo Mini Cognitive Exam (MEC),
* Those people who due to their physical condition cannot carry out the tests with guarantees of safety.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active people over 60 years of age recruited from two associations from the city of Valencia, Spain will be part of the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Health status | day 1
  By the SF-12 Health Questionnaire (version 2). This questionnaire is an abbreviated version of the SF-36, with an approximate duration of 2 minutes and made up of 12 different items that address different physical and mental aspects of the person (physical role, emotional role, social role, physical function, mental health , limiting pain, vitality and general health). It uses the Likert scale and each item has different response options ranging from 3 to 6. The maximum score that can be obtained is 100 points.

SECONDARY OUTCOMES:
Intensity of Pain | day 1
  Visual Analog Scale. It is a commonly used and validated instrument in the interpretation of pain intensity. In a line of 10 cm, divided by numbers from 0 to 10, the patient marks the intensity of the pain, being 0 "absence of pain" and 10 "worst pain imaginable".
Mental State | day 1
  By Minimental State Examination. It is made up of a set of items that are grouped into 5 groups or cognitive areas: orientation in space and time (2 items), fixation (1 item), concentration and calculation (2 items), memory (1 item), and language and construction (7 items). Throughout its completion it is important to speak clearly to the participants and in the event of a mistake not to correct them and to continue with the questionnaire. Each item is evaluated from 0 to 5, with 5 being the maximum score that can be achieved when the question is answered correctly. The maximum score of the exam is 35 points, being normal values: between 30 and 35 and indicating cognitive impairment scores below 24 (in people over 65) and below 28 (in people 65 years or less)
Level of Physical Activity | day 1
  Physical activity was measured by the Short Form-International Physical Activity Questionnaire (s-IPAQ). The s-IPAQ contains seven items for identifying the frequency and duration of light, moderate, and vigorous physical activity as well as inactivity during the past week. The questions focus on four activity types: "vigorous activity" periods of at least 10 minutes, "moderate activity" periods of at least 10 minutes, "walking" periods of at least 10 minutes, and times spent "sitting" on weekdays. Frequency of activity is measured in days, and duration in hours and minutes. The patients were classified into three physical activity categories: low, moderate, and high. Typical s-IPAQ correlations with an accelerometer were 0.80 for reliability.
Sleep quality | day 1
  Using the Pittsburg questionnaire (ICSP). It consists of 19 items or questions from which an overall score is obtained and which in turn are grouped into 7 different components (subjective sleep quality, latency, duration, sleep efficiency, sleep disturbances, use of medication and daytime dysfunction) . The total score will range from 0 to 21, with a higher score signifying a serious sleep problem. Values less than 5 indicate normality, values between 5 and 7 suggest medical attention, between 8 and 14 would be adequate medical attention and treatment, and a score greater than 15 is significant for a serious sleep problem.
Mood State | day 1
  Goldberg depression and anxiety. It is a questionnaire that presents two scales, one for depression and the other for anxiety. Each one of these is made up of 4 initial items or questions to test and determine if there is a probability of the presence of one of these disorders, and another 5 items that are only formulated if the patient has answered affirmatively in the first 4. On the one hand, in the anxiety scale, the question is continued in the case of 2 or more affirmative answers in the first 4 questions, and in the depression scale, the questions are continued if there is any affirmative answer in the first 4 items. Regarding the final score, on the anxiety scale, 4 or more affirmative answers probably indicate an anxiety disorder, and on the depression scale 2 or more positive answers indicate a possible depressive disorder.
Exercise tolerance | day 1
  6 Six Minute Walk Test (6MWT). The object of this test is to walk as far as possible for 6 minutes. The patient will walk back and forth around the cones in a hallway and is permitted to slow down, to stop, and to rest as necessary (but resume walking as soon as able)
Forced spirometry | day 1
  Assessed using a COSMED PONY FX spirometer with mouthpiece and filters (1 cardboard mouthpiece and a bacteriological filter per patient). The test was performed with the person sitting, without crossing the legs and shoulders relaxed. Anthropometric data were entered into the equipment, nose was covered with a nose clio and the patient was then asked to perform three forced inhalations and exhalations.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí López, Dr, Principal Investigator — University of Valencia
Locations (1):
- Gemma Victoria Espí-López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No